CLINICAL TRIAL: NCT04657601
Title: Prospective Evaluation Utilizing an Endolumenal Interventional Platform Device to Facilitate Endoscopic Polypectomy
Brief Title: Prospective Study of a New Endolumenal Device Used During Endoscopic Polypectomy in the Colon
Acronym: DiLumenC2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lumendi, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: USLUM 1802 or 2020-01
Record Dates: First submitted 2020-10-22; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Polyps of Colon
Keywords: Intestinal Polyps; Pathologic Condition, Anatomical; Polyps
MeSH Terms: conditions — Colonic Polyps; Intestinal Polyps; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Patients undergo polypectomy facilitated by the study device.
  Interventions: Device: DiLumen C2 Endolumenal Interventional Platform

INTERVENTIONS:
Device: DiLumen C2 Endolumenal Interventional Platform — Dual balloon accessory to an endoscope and related instruments

SUMMARY:
This prospective observational study will evaluate the performance of the DiLumen C2 Endolumenal Interventional Platform and its instruments. Up to 100 subjects will be enrolled at up to 5 clinical sites. Patient data will be collected before the procedure, during the procedure, and up until the patient is discharged from the hospital.

DETAILED DESCRIPTION:
This study is a prospective, post-market evaluation of the performance of the DiLumen C2 Endolumenal Interventional Platform ("C2 device") used as an endoscopic dual balloon accessory device used to ensure complete positioning, visualization, and diagnosis in endoscopic treatments in the large intestine. The DiLumen Endolumenal Interventional Knife ("IK device") and the DiLumen Endolumenal Interventional Grasper ("IG device") are disposable instruments used with the C2 device. These devices are cleared by the US Food and Drug Administration (FDA) for commercial use in endolumenal therapies and will be used on-label in this study. The overall goal of this study is to evaluate the clinical performance of the C2 device and its related instruments. Intra-procedure parameters (procedure timepoints, anesthesia use, polyp location and description), final pathology/histology, and general complications will also be evaluated. Investigators will also be asked to assess the ease of use of the C2Interventional Platform.

To accomplish this goal, up to 100 subjects will be enrolled at up to 5 clinical sites and treated using the C2 device and related instruments. Evaluations will be performed pre-procedure, during the procedure, and at discharge. Assessments will include polyp classification/pathology, procedure timepoints, final pathology/histology, adverse events, and ease of use. As per the FDA cleared product labeling this study will be limited to subjects undergoing an endoscopic procedure to remove polyps in the large intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18-85 years of age.
2. Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Scheduled for endoscopic removal of suspected colorectal adenomatous polyps which are sessile or polypoid lesions.
4. Have, in the opinion of the Investigator(s) or co-investigator(s), no medical contraindication to endoscopic submucosal dissection (ESD).

Exclusion Criteria:

1. Have a contraindication to colonoscopy, including but not limited to active colitis, diverticulitis, perforation, or stricture.
2. Have a history of open or laparoscopic colorectal surgery.
3. Have a history of Inflammatory Bowel Disease (IBD).
4. Have a suspected invasive malignancy on polyp assessment.
5. Any medical or surgical condition that would preclude the potential benefit ESD.
6. Any case where the device or instrument would be too large or too small to achieve a successful result.
7. Anatomy or other factors that prohibit safe access to the large intestine such as previous radiation therapy to the affected area.
8. History of AIDS, HIV, or active hepatitis.
9. History of mental illness, including psychological or neurological conditions (addiction to substances such as alcohol. e.g.) that in the investigator's opinion would pre-empt their ability or willingness to participate in the study.
10. Has cardiopulmonary conditions that present prohibitive anesthesia risk.
11. Has uncorrectable coagulopathy or hemorrhagic diathesis.
12. Has an active infection or fever.
13. Has allergy to any component of the treatment procedure.
14. Patients who are pregnant.
15. Pediatric case (Age < 18 years)
16. Any case in which use of the DiLumen C2 device is not needed.
17. Any case not described in the indications.
18. Currently involved in another investigational product for similar purposes.
19. Prisoners.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population includes adults (ages 18-85 years) men and women scheduled to undergo a colorectal ESD. Subjects will be recruited from the investigator's standard patient population as seen in their routine clinical practice and will be screened for participation according to the protocol defined inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The ability of the investigator to perform an endoscopic ESD safely and effectively | Through study completion, up to 7 days
  Whether or not the polyp was removed and if there were any adverse events

SECONDARY OUTCOMES:
Details of the procedure | Through study completion, up to 7 days
  Procedure time
Details of the procedure | Through study completion, up to 7 days
  Dissection speed
Legnth of Hospital Stay | Through study completion, up to 7 days
  How long the patient was in the hospital following the polypectomy